CLINICAL TRIAL: NCT00521144
Title: Phase I/II Study of Obatoclax Mesylate (GX15-070MS), a Bcl-2 Antagonist, Plus Topotecan in Relapsed Small Cell Lung Carcinoma
Brief Title: Obatoclax Mesylate and Topotecan Hydrochloride in Treating Patients With Relapsed or Refractory Small Cell Lung Cancer or Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00252; 07-082 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000561779 (Registry Identifier: PDQ (Physician Data Query)); NCT01645657 (obsolete NCT alias)
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Results first posted 2014-07-22 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2013-12

CONDITIONS: Recurrent Small Cell Lung Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — obatoclax; Topotecan; trioctyl phosphine oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor therapy and chemotherapy) (Experimental): Patients receive obatoclax mesylate IV over 3 hours on day 1 OR days 1 and 3 and topotecan hydrochloride IV over 30 minutes on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: obatoclax mesylate; Drug: topotecan hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: obatoclax mesylate — Given IV
  Other Names: GX15-070MS
Drug: topotecan hydrochloride — Given IV
  Other Names: hycamptamine; Hycamtin; SKF S-104864-A; TOPO
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I/II trial is studying the side effects and best dose of obatoclax mesylate when given together with topotecan hydrochloride and to see how well they work in treating patients with relapsed or refractory small cell lung cancer or advanced solid tumors. Obatoclax mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as topotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving obatoclax mesylate together with topotecan hydrochloride may help kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose, recommended phase II dose, and toxicity profile of obatoclax mesylate when administered with topotecan hydrochloride in patients with advanced solid tumors. (Phase I) II. Determine the response rate in patients with relapsed or refractory small cell lung cancer treated with obatoclax mesylate and topotecan hydrochloride. (Phase II)

SECONDARY OBJECTIVES:

I. Evaluate the expression of pro- and anti-apoptotic proteins which may correlate with obatoclax mesylate sensitivity or resistance.

OUTLINE: This is a phase I dose-escalation study of obatoclax mesylate followed by a phase II study.

PHASE I (solid tumor): Patients receive obatoclax mesylate IV over 3 hours on day 1 OR days 1 and 3 and topotecan hydrochloride IV over 30 minutes on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

PHASE II (small cell lung cancer): Patients receive obatoclax mesylate and topotecan hydrochloride at the recommended phase II dose (RPTD) determined in phase I. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Tumor tissue samples from patients with small cell lung cancer may be collected at baseline for correlative studies. Tissue samples are analyzed for biomarkers and protein expression of Bcl-2, Bcl-Xl, MCL-1, Bax, Bad, c-Myc, L-Myc, and N-Myc by immunohistochemistry.

After completion of study treatment, patients are followed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of 1 of the following:

  * Advanced solid tumor (phase I)

    * Topotecan hydrochloride must be an appropriate treatment for this cancer
  * Small cell lung cancer (SCLC) (phase II)

    * Progressed after one prior platinum-based chemotherapy regimen
    * Pathology materials (tumor tissue) will be used for correlative studies, if available
* No progressive brain metastases

  * Treated brain metastases allowed provided patient is neurologically stable and does not require steroids
* No leptomeningeal involvement
* ECOG performance status (PS) 0-1 OR Karnofsky PS 70-100%
* Leukocytes ≥ 3,000/mcL
* Absolute neutrophil count ≥ 1,500/mcL
* Platelet count ≥ 100,000/mcL
* Total bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Fertile patients must use effective double barrier method of contraception during and for 3 months after completion of study therapy
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents or anticancer therapy

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biological composition to obatoclax mesylate or topotecan hydrochloride (e.g., irinotecan)
* Concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would limit compliance with study requirements
* History of seizure disorder or other neurological dysfunction (except peripheral neuropathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Krug, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Paik PK, Rudin CM, Pietanza MC, Brown A, Rizvi NA, Takebe N, Travis W, James L, Ginsberg MS, Juergens R, Markus S, Tyson L, Subzwari S, Kris MG, Krug LM. A phase II study of obatoclax mesylate, a Bcl-2 antagonist, plus topotecan in relapsed small cell lung cancer. Lung Cancer. 2011 Dec;74(3):481-5. doi: 10.1016/j.lungcan.2011.05.005. Epub 2011 May 26. PMID 21620511

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 8/7/2007 Primary Completion Date 8/10/2010 Recruitment Location at medical clinic
Groups:
- Phase I; Level 1: Obatoclax Mesylate + Topetecan: Level 1: Obatoclax Mesylate (GX15-070MS) 3 hour infusion, days 1 (and 3), q21 days, 14 mg/m2: Topotecan days 1-5, q21 days, 1.25 mg/m2
- Phase I; Level 2: Obatoclax Mesylate + Topetecan: Level 2: Obatoclax Mesylate (GX15-070MS) 3 hour infusion, days 1 (and 3), q21 days, 20 mg/m2: Topotecan days 1-5, q21 days, 1.25 mg/m2
- Phase I; Level 3: Obatoclax Mesylate + Topetecan: Level 3: Obatoclax Mesylate (GX15-070MS) 3 hour infusion, days 1 (and 3), q21 days, 14 + 14 mg/m2: Topotecan days 1-5, q21 days, 1.25 mg/m2
- Phase I; Level 4: Obatoclax Mesylate + Topotecan: Level 4: Obatoclax Mesylate (GX15-070MS) 3 hour infusion, days 1 (and 3), q21 days, 20 + 20 mg/m2: Topotecan days 1-5, q21 days, 1.25 mg/m2
- Phase II Obatoclax Mesylate + Topotecan in SCLC: Obatoclax Mesylate 14 + 14 mg/m2 and Topotecan 1.25 mg/m2
Period: Overall Study
Arm/Group | Phase I; Level 1: Obatoclax Mesylate + Topetecan | Phase I; Level 2: Obatoclax Mesylate + Topetecan | Phase I; Level 3: Obatoclax Mesylate + Topetecan | Phase I; Level 4: Obatoclax Mesylate + Topotecan | Phase II Obatoclax Mesylate + Topotecan in SCLC
Started | 6 | 5 | 3 | 1 | 7
Completed | 2 | 2 | 1 | 0 | 0
Not Completed | 4 | 3 | 2 | 1 | 7
Not completed — Not Treated | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 1
Not completed — Progressive Disease | 4 | 2 | 2 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Phase I Obatoclax Mesylate + Topotecan in Solid Tumors Level 1: Level 1: Obatoclax Mesylate (GX15-070MS) 3 hour infusion, days 1 (and 3), q21 days, 14 mg/m2: Topotecan days 1-5, q21 days, 1.25 mg/m2
- Phase I Obatoclax Mesylate + Topotecan in Solid Tumors Level 2: Level 2: Obatoclax Mesylate (GX15-070MS) 3 hour infusion, days 1 (and 3), q21 days, 20 mg/m2: Topotecan days 1-5, q21 days, 1.25 mg/m2
- Phase I Obatoclax Mesylate + Topotecan in Solid Tumors Level 3: Level 3: Obatoclax Mesylate (GX15-070MS) 3 hour infusion, days 1 (and 3), q21 days, 14 + 14 mg/m2: Topotecan days 1-5, q21 days, 1.25 mg/m2
- Phase I Obatoclax Mesylate + Topotecan in Solid Tumors Level 4: Level 4: Obatoclax Mesylate (GX15-070MS) 3 hour infusion, days 1 (and 3), q21 days, 20 + 20 mg/m2: Topotecan days 1-5, q21 days, 1.25 mg/m2
- Total: Total of all reporting groups
Arm/Group | Phase I Obatoclax Mesylate + Topotecan in Solid Tumors Level 1 | Phase I Obatoclax Mesylate + Topotecan in Solid Tumors Level 2 | Phase I Obatoclax Mesylate + Topotecan in Solid Tumors Level 3 | Phase I Obatoclax Mesylate + Topotecan in Solid Tumors Level 4 | Phase II Obatoclax Mesylate + Topotecan in SCLC | Total
Number analyzed (Participants) | 6 | 5 | 3 | 1 | 7 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 2 | 0 | 4 | 14
  >=65 years | 1 | 2 | 1 | 1 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 1 | 1 | 6 | 14
  Male | 1 | 4 | 2 | 0 | 1 | 8
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 3 | 1 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Phase II)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR)=CR +PR
Time Frame: Every 6 weeks, assessed up to 30 days
Population: Only those patients who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response.
Measure: Number; unit: participants
Groups:
- Phase 1; Level 4: Obatoclax Mesylate + Topotecan: Obatoclax Mesylate (GX15-070MS) 3 hour infusion, days 1 (and 3), q21 days, 20 + 20 mg/m2: Topotecan days 1-5, q21 days, 1.25 mg/m2
Arm/Group | Phase I; Level 1: Obatoclax Mesylate + Topetecan | Phase I; Level 2: Obatoclax Mesylate + Topetecan | Phase I; Level 3: Obatoclax Mesylate + Topetecan | Phase 1; Level 4: Obatoclax Mesylate + Topotecan | Phase II Obatoclax Mesylate + Topotecan in SCLC
Number analyzed (Participants) | 6 | 5 | 3 | 0 | 7
participants | 0 | 0 | 0 |  | 0

ADVERSE EVENTS:
Groups:
- Phase I; Level 1: Obatoclax Mesylate + Topotecan: Level 1: Obatoclax Mesylate (GX15-070MS) 3 hour infusion, days 1 (and 3), q21 days, 14 mg/m2: Topotecan days 1-5, q21 days, 1.25 mg/m2
- Phase I; Level 2: Obatoclax Mesylate + Topotecan: Level 2: Obatoclax Mesylate (GX15-070MS) 3 hour infusion, days 1 (and 3), q21 days, 20 mg/m2: Topotecan days 1-5, q21 days, 1.25 mg/m2
- Phase I; Level 3: Obatoclax Mesylate + Topotecan: Level 3: Obatoclax Mesylate (GX15-070MS) 3 hour infusion, days 1 (and 3), q21 days, 14 + 14 mg/m2: Topotecan days 1-5, q21 days, 1.25 mg/m2
Arm/Group | Phase I; Level 1: Obatoclax Mesylate + Topotecan | Phase I; Level 2: Obatoclax Mesylate + Topotecan | Phase I; Level 3: Obatoclax Mesylate + Topotecan | Phase I; Level 4: Obatoclax Mesylate + Topotecan | Phase II Obatoclax Mesylate + Topotecan in SCLC
Serious Adverse Events (participants affected / at risk) | 4/6 | 4/5 | 2/3 | 0/1 | 4/7
Other Adverse Events (participants affected / at risk) | 6/6 | 3/5 | 2/3 | 0/1 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I; Level 1: Obatoclax Mesylate + Topotecan (N=6) | Phase I; Level 2: Obatoclax Mesylate + Topotecan (N=5) | Phase I; Level 3: Obatoclax Mesylate + Topotecan (N=3) | Phase I; Level 4: Obatoclax Mesylate + Topotecan (N=1) | Phase II Obatoclax Mesylate + Topotecan in SCLC (N=7)
Ataxia (incoordination) (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Euphoria (Psychiatric disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anemia-Hemoglobin decrease (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Allergic Reaction-Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALT, SGPT (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alkaline phosphatase (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
AST, SGOT (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Blood bilirubin increase (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesemia (low magnesium) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death-NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infection, other (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I; Level 1: Obatoclax Mesylate + Topotecan (N=6) | Phase I; Level 2: Obatoclax Mesylate + Topotecan (N=5) | Phase I; Level 3: Obatoclax Mesylate + Topotecan (N=3) | Phase I; Level 4: Obatoclax Mesylate + Topotecan (N=1) | Phase II Obatoclax Mesylate + Topotecan in SCLC (N=7)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ataxia (incoordination) (Nervous system disorders) | 5 (11) | 2 (6) | 2 (4) | 0 (0) | 7 (21)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (6)
Fatigue (General disorders) | 4 (6) | 2 (4) | 2 (3) | 0 (0) | 5 (7)
Glomerular filtration rate decrease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anemia-Hemoglobin decrease (Metabolism and nutrition disorders) | 3 (6) | 2 (2) | 0 (0) | 0 (0) | 4 (22)
Hemorrhage, Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (3)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decrease (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 6 (14)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Euphoria (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis-oral (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (6) | 2 (4) | 1 (1) | 0 (0) | 3 (6)
Neutrophil count decrease (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (7)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decrease (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 6 (16)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 4 (7) | 3 (6) | 1 (1) | 0 (0) | 7 (31)
Dysgeusia (taste alteration) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Speech impairment (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALT, SGPT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
AST, SGOT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Alkaline phosphatase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (8)
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Mucosal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decrease (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mood alteration-Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy-sensory (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pain-Head/Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less